CLINICAL TRIAL: NCT01212328
Title: Developing and Testing Integrated, Multi-factorial Cardiovascular Disease Risk Reduction Strategies in South Asia (CARRS Translation Trial)
Brief Title: A Multi-site, Individually Randomized, Controlled Translation Trial of Integrated and Comprehensive Care Strategies to Reduce Cardiovascular Disease (CVD) Risk Among 1,120 Type 2 Diabetes Mellitus(T2DM) Patients in South Asia
Acronym: CARRS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Public Health Foundation of India (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH); United Health Group, USA (Unknown); All India Institute of Medical Sciences (Other); Madras Diabetes Research Foundation, Chennai (Unknown); Aga Khan University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: UTRN 022342347-29072010248
Record Dates: First submitted 2010-09-06; First posted 2010-09-30 (Estimated); Last update posted 2011-09-05 (Estimated); Status verified 2011-09

CONDITIONS: Type 2 Diabetes Mellitus; Hypertension; Dyslipidaemia
Keywords: T2DM; Decision support software; care coordinator
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Hypertension; Dyslipidemias

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Care coordinator + Decision Support Software (Experimental): Care coordinator + Decision Support Software (Experimental Arm): The patients will receive integrated diabetes care management consisting of current diabetes management guidelines + Non-Physician care coordinator assistance + Electronic Health Records- Decision Support Software (EHR-DSS) (The software will generate diabetes management prompts for the treating physician and reminders for clinic visits for the intervention arm patients.)
  Interventions: Other: Care Coordinator + Decision Support Software
- Usual care (Active Comparator): Usual care (Active Comparator Arm): Patients will continue with the usual diabetes care with no care coordinator assistance and no decision support software - management prompt.
  Interventions: Other: Usual care

INTERVENTIONS:
Other: Care Coordinator + Decision Support Software — Care coordinator + Decision Support Software (Experimental Arm): The patients will receive integrated diabetes care management consisting of current diabetes management guidelines + Non-Physician care coordinator assistance + Electronic Health Records- Decision Support Software (EHR-DSS) (The software will generate diabetes management prompts for the treating physician and reminders for clinic visits for the intervention arm patients.)
  Arms: Care coordinator + Decision Support Software
Other: Usual care — Usual care (Active Comparator Arm): Patients will continue with the usual diabetes care with no care coordinator assistance and no decision support software - management prompt.
  Arms: Usual care

SUMMARY:
Background: Cardiovascular diseases (CVD) are currently the leading cause of death globally and Asian Indians will account for between 40-60% of the global CVD burden within the next 10-15 years. Risk factor control and preventive care are effective in reducing CVD events and mortality. The greatest gains in CVD prevention have been seen when early and target-driven interventions address multiple risk factors together. However, achieving control of even individual risk factors (blood glucose, blood pressure, or blood lipid targets) is poor, globally. Quality improvement schemes, like the proposed intervention, have shown promise in high-income countries, but are untested in South Asia; a region with a population at extraordinarily high CVD risk.

Objective: To test whether a clinic-based case management intervention (consisting of guidelines based treatment, care coordinator assistance and decision support software) to reduce cardiovascular disease (CVD) risk among Type 2 diabetes patients in South Asia, is more effective and sustainable compared to existing care.

Trial subjects and methods: The study will involve a total of 1120 patients attending 8 established out-patient clinics in South Asia (140 patients at each clinic). Patients enrolled in the trial will be randomly assigned to either the control (existing care) or the intervention group and will be followed up for an average of 30 months. The total trial duration is about 3.5 years, from mid-August 2010 to December 31, 2013.

ELIGIBILITY:
Inclusion Criteria:

1. Age 35 years and older
2. Confirmed diagnosis of diabetes based on documented evidence from oral glucose tolerance test or two venous fasting blood sugar levels or known diabetes patient on medication or insulin
3. Poor glycemic control (as evidenced by HbA1c >=8.0%) and one or both of: dyslipidemia [Low density Lipoprotein (LDL) >=130 mg/dl] or systolic hypertension [Systolic Blood Pressure (SBP) >=140 mmHg], irrespective of lipid- or BP-lowering medication use, respectively
4. Receiving diabetes care in the same clinic for at least 3 months OR even earlier if in the investigator's assessment the patient is likely to follow-up regularly as required by the protocol.
5. Willingness to consent to randomization.

Exclusion Criteria:

Individuals will be excluded from participation if any of the following are present during screening:

1. Known type 1 diabetes mellitus
2. Diabetes secondary to chronic pancreatitis
3. Pregnant OR trying to become pregnant OR of child-bearing potential and not actively practicing birth control (including natural methods)
4. Evidence of pre-existing well-controlled blood glucose, blood pressure or LDL-cholesterol (as evidenced by HbA1c < 7.0%, SBP < 130 mmHg, LDL-cholesterol < 100 mg/dl [LDL-cholesterol < 70 mg/dl with history of CVD event]) obtained from screening within a period not exceeding 28 days (4 weeks) prior to randomization
5. Documented cardiovascular event (coronary revascularization, stroke, MI, unstable angina) in past 12 months
6. Current symptomatic Congestive Heart Failure (CHF) or New York Heart Association (NYHA) Class 3 or 4 effort intolerance
7. Documented non-diabetic kidney disease OR pre-existing end -stage renal disease (on renal replacement therapy [dialysis or transplant])
8. Transaminase >3 times upper limit of normal OR active liver disease within past 2 years
9. Malignancy or life-threatening disease with death probable in 4 years
10. Any current medication (e.g. long-term steroids, protease inhibitors) that, in the opinion of the site investigator, would interfere with participant's diabetic status and follow-up
11. Any condition or circumstance that is unrelated to diabetes progression, that in the opinion of the site investigator would interfere with the participant's diabetic status and follow-up: including (but not limited to) other endocrinopathy [adrenal, pituitary], Tuberculosis (TB) patient on treatment, psychiatric illness or cognitive impairment, alcohol or drug abuse, history of organ transplant, Body Mass index (BMI) >= 45 kg/m2
12. On an investigational drug in the last 3 months
13. Currently participating in a clinical trial
14. No fixed address or contact details
15. Plans to move in the next 3 years
16. A member of the participant's household is currently in the trial
17. Inability or unwillingness of individual or legal guardian /representative to give written informed consent

Min Age: 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1120 (Estimated)
Dates: Start 2010-10; Primary Completion 2013-12 (Estimated); Study Completion 2014-06 (Estimated)

PRIMARY OUTCOMES:
Multiple CVD risk factor control targets | 42 months after randomization
  The study has one primary outcome of interest, multiple CVD risk factor control targets: at least two targets including Hemoglobin A1c (HbA1c) < 7.0% and at least one of: Blood Pressure (BP) < 130/80 mmHg or Low Density Lipoprotein (LDL)-cholesterol < 100 mg/dl (LDL cholesterol < 70 mg/dl for those with history of CVD event)

SECONDARY OUTCOMES:
Single risk factor control of at least one target either HbA1c or blood pressure or LDL-Cholesterol | 42 months after randomization
  Single risk factor control
  1. absolute 10% point greater proportion of participants in the intervention group achieving good glycemic control (HbA1c < 7%)
  2. systolic BP < 130 and diastolic BP < 80 mmHg
  3. LDL-cholesterol < 100 mg/dl, < 70 mg/dl for those with history of CVD event)
The cost effectiveness analysis of the intervention compared to the usual care. | 42 months after randomization
Quality of life | 42 months after randomization
Prescriber and patient acceptability of the Digital Support software and care coordinator with management guidelines. | 42 months after randomization

CONTACTS AND LOCATIONS:
Overall Officials: Dorairaj Prabhakaran, MD, DM, MSc., Principal Investigator — Public Health Foundation of India
Locations (10):
- India (9):
  - Bangalore Endocrinology and Diabetes Research Centre,, #35, 5th Cross,Malleswaram Circle,, Bangalore, Karnataka
  - St. John's Medical College & Hospital,, Sarjapur Road, Koramangala,, Bangalore
  - Diabetes Research Centre & MV Hospital for Diabetes,, No 4 West Madha Church Street, Royapuram, Chennai
  - Endocrine Division, Department of Medicine, Goa Medical College,, Bambolim, Goa
  - Department of Endocrinology, CARE Hospital,, Road No 1, Banjara Hills,, Hyderabad,
  - Osmania General Hospital,, 2nd Floor, Golden Jubilee Block, Afzalgunj,, Hyderabad
  - Amrita Institute of Medical Sciences, Kochi, Kerala
  - Topiwala National Medical College & BYL Nair Ch. Hospital,, Dr. A. L. Nair Road, Mumbai Central,, Mumbai
  - Public Health Foundation of India, New Delhi, National Capital Territory of Delhi
- Department of CHS, The Aga Khan, University,, P.O. BOx. 3500 Stadium, Road,, Karachi, Pakistan

REFERENCES:
- [Derived] Cashmore BA, Cooper TE, Evangelidis NM, Green SC, Lopez-Vargas P, Tunnicliffe DJ. Education programmes for people with chronic kidney disease and diabetes. Cochrane Database Syst Rev. 2024 Aug 22;8(8):CD007374. doi: 10.1002/14651858.CD007374.pub3. PMID 39171639
- [Derived] Singh K, Kondal D, Jagannathan R, Ali MK, Prabhakaran D, Narayan KMV, Anand S, Tandon N; CARRS Trial Investigators. Rate and risk factors of kidney function decline among South Asians with type 2 diabetes: analysis of the CARRS Trial. BMJ Open Diabetes Res Care. 2024 Aug 16;12(4):e004218. doi: 10.1136/bmjdrc-2024-004218. PMID 39153754
- [Derived] Ali MK, Singh K, Kondal D, Devarajan R, Patel SA, Menon VU, Varthakavi PK, Vishwanathan V, Dharmalingam M, Bantwal G, Sahay RK, Masood MQ, Khadgawat R, Desai A, Prabhakaran D, Narayan KMV, Tandon N. Effect of a multicomponent quality improvement strategy on sustained achievement of diabetes care goals and macrovascular and microvascular complications in South Asia at 6.5 years follow-up: Post hoc analyses of the CARRS randomized clinical trial. PLoS Med. 2024 Jun 3;21(6):e1004335. doi: 10.1371/journal.pmed.1004335. eCollection 2024 Jun. PMID 38829880
- [Derived] Singh K, Ali MK, Devarajan R, Shivashankar R, Kondal D, Ajay VS, Menon VU, Varthakavi PK, Viswanathan V, Dharmalingam M, Bantwal G, Sahay RK, Masood MQ, Khadgawat R, Desai A, Prabhakaran D, Narayan KMV, Phillips VL, Tandon N; CARRS Trial Group. Rationale and protocol for estimating the economic value of a multicomponent quality improvement strategy for diabetes care in South Asia. Glob Health Res Policy. 2019 Mar 18;4:7. doi: 10.1186/s41256-019-0099-x. eCollection 2019. PMID 30923749
- [Derived] Ali MK, Singh K, Kondal D, Devarajan R, Patel SA, Shivashankar R, Ajay VS, Unnikrishnan AG, Menon VU, Varthakavi PK, Viswanathan V, Dharmalingam M, Bantwal G, Sahay RK, Masood MQ, Khadgawat R, Desai A, Sethi B, Prabhakaran D, Narayan KM, Tandon N; CARRS Trial Group. Effectiveness of a Multicomponent Quality Improvement Strategy to Improve Achievement of Diabetes Care Goals: A Randomized, Controlled Trial. Ann Intern Med. 2016 Sep 20;165(6):399-408. doi: 10.7326/M15-2807. Epub 2016 Jul 12. PMID 27398874
- [Derived] CARRS Trial Writing Group; Shah S, Singh K, Ali MK, Mohan V, Kadir MM, Unnikrishnan AG, Sahay RK, Varthakavi P, Dharmalingam M, Viswanathan V, Masood Q, Bantwal G, Khadgawat R, Desai A, Sethi BK, Shivashankar R, Ajay VS, Reddy KS, Narayan KM, Prabhakaran D, Tandon N. Improving diabetes care: multi-component cardiovascular disease risk reduction strategies for people with diabetes in South Asia--the CARRS multi-center translation trial. Diabetes Res Clin Pract. 2012 Nov;98(2):285-94. doi: 10.1016/j.diabres.2012.09.023. Epub 2012 Oct 22. PMID 23084280